CLINICAL TRIAL: NCT07035600
Title: WASA - Walking and Sitting Difficulties After APE
Brief Title: Walking and Sitting Difficulties After Rectal Cancer Surgery
Acronym: WASA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Principal Investigator, Charlotta Larsson, MD PhD, MD PhD, Göteborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2024-08611-01
Record Dates: First submitted 2025-04-08; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Rectal Cancer Patients; Rectal Cancer Surgery; Rectal Cancer, Radiotherapy; Rectal Cancer
Keywords: Rectal cancer; Rectal cancer complications
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized, interventional, controlled mtrial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training intervention arm (Experimental): Targeted supervised training program of specific training of levator, abdominal, quadriceps (all portions), and gluteal muscles as well as endurance training.
  Interventions: Procedure: Targeted leaderled training program
- Control arm (Active Comparator): Information of training in accordance with WHO recommendations of 30 min aerobic physical activity five times per week (150 min per week) plus strength sessions twice weekly.
  Interventions: Procedure: Control arm with WHO recommendation on physical activity

INTERVENTIONS:
Procedure: Targeted leaderled training program — Training program:
  After inclusion and consent the patients are instructed through an online group training program consisting of specific training of levator, abdominal, quadriceps (all portions), and gluteal muscles as well as endurance training. They are given information about WHO recommendations about physical activity. The patients are asked to sign up for two specific training occasions per week where no group will be larger than 10 patients. Group based exercise sessions consist of 45-minute supervised online zoom exercise sessions. Apart from the supervised sessions patients are encouraged to perform one functional training session, unsupervised, as well as follow the WHO recommendation for aerobic exercise
  Arms: Training intervention arm
Procedure: Control arm with WHO recommendation on physical activity — Training will be in accordance with WHO recommendations of 30 min aerobic physical activity five times per week (150 min per week) plus strength sessions twice weekly. The patients will be individually adviced on how to perform the training at inclusion in the trial. This is considered standard care and will not include any on-line supervision, but will include a coaching/reminder by a phone call from a research nurse/short message service (by choice of the patient) at regular intervals before and after surgery
  Arms: Control arm

SUMMARY:
Earlier studies have shown that many patients (up to 30%) who have had a major surgery for rectal cancer, called a rectum amputation (where the entire rectum and anus are removed and the person gets a permanent stoma), still have trouble sitting and walking three years after the surgery. These problems are then seen as long-term or chronic.

WASA is a randomized multicenter international study that will test a way to reduce these problems. It will start in fall 2025 and go on for 3.5 years. About 300 patients will take part.

The patients will be randomly divided into two groups. One group will get guided online training twice a week, specially made for their needs. The other group will get information about the World Health Organization's (WHO) general advice on physical activity.

The idea is that special training during the first year after surgery will reduce problems with walking and sitting. If the hypothesis can be confirmed, it could lead to an easy and low-cost way to help many rectal cancer patients feel and function better.

DETAILED DESCRIPTION:
Coordinating centre:

SSORG/Göteborg, Department of Surgery, Sahlgrenska University Hospital/Östra Principal Investigator: Charlotta Larsson MD, PhD Deputy Principal Investigator: Eva Haglind, MD, PhD, professor emerita Doctoral student: Lina Björklund Sand MD

Purpose and Aims:

The primary aim of the WASA trial is to evaluate the effectiveness of a structured physical activity program compared to standard WHO-based physical activity recommendations in reducing sitting and walking difficulties in patients who have undergone abdominoperineal excision (APE) for rectal cancer. The intervention secondary aims are to improve patient quality of life and reduce chronic pain and mobility issues post-surgery.

Background:

Surgery is the mainstay for curative treatment of the vast majority of rectal cancers, often in combination with chemoradiotherapy before the operation. For low rectal cancer abdominoperineal excision (APE) is performed, in cases with tumour involvement of the levators, including part/all of the levators in the removed specimen (ELAPE). In extralevator abdominoperineal excision (ELAPE) reconstruction of the pelvic floor is part of the procedure. All patients will have a permanent stoma.

In a national cohort of Swedish patients who had undergone APE/ELAPE during 2011 -2013 questionnaires distributed 3 years postoperatively and based on themes that occurred during semi-structured interviews before construction of the questionnaire, included questions about sitting and walking difficulties as well as pain. In the analyses we found that 20-25% of patients experienced sitting and/or walking difficulties, and/or pain, which thus should be regarded as chronic (1). In a multicentre, international and prospective study of patients with rectal cancer, we found that up to 30% of patients had sitting and/or walking difficulties 2 years after APE and that significantly fewer patients who had been operated by an anterior resection experienced such problems (2).

Few if any other reports have focused on these problems, which could lead to impairments of normal daily living.

The aim of this trial is to compare the effect an intervention consisting of a specific program of physical activity introduced before surgery and continued for 12 months after surgery in comparison with a control group receiving information about physical activity as recommended by WHO.

The underlaying hypothesis is that by increasing muscle mass and -strength in muscle groups in the pelvis, lower abdominal and upper thigh area as well as balance training the difficulties in sitting and walking after abdominoperineal excision will decrease.

Study plan, preliminary results and clinical relevance

Study design

The design is randomized, international, multicentre comparing an intervention consisting of a specific, supervised live online training program introduced after diagnosis and before surgery/neoadjuvant treatment with adaptions immediately after surgery (index surgery) with a control group where patients are carefully informed of the physical activity as recommended by WHO. The design involves all consecutive, consenting patients with rectal cancer to be treated by APE with/without neoadjuvant treatment in participating hospitals.

The randomization will be stratified by ELAPE/APE, hospital and neoadjuvant treatment.

Patients will be accrued from the hospitals within the SSORG network and consenting to participate in the trial after information. Other surgical departments with interest are welcome to join in the trial. Patients will undergo surgery, follow-up and adjuvant treatment according to local routine.

Training program

Intervention group After inclusion and consent the patients are instructed trough an online leader-led group training program consisting of specific training of mainly levator, abdominal, quadriceps (all portions) and gluteal muscles as well as endurance training. They are given information about WHO recommendation about physical activity. The patients are asked to sign up for two specific training sessions per week. Group size maximum 10 patients.

Control group After inclusion careful instruction about WHO recommendations on physical activity with 30 min aerobic physical activity 5 times per week/150 min per week plus strength sessions twice weekly.

Outcome Measures

* Primary Outcome: Measurement of self-reported sitting and walking difficulties at 12 months post-surgery.
* Secondary Outcomes: Measurement of self-reported sitting and walking difficulties at 6 and 24 months post-surgery, objective measures including a 6-minute walking test and standardized balance tests, complications, patient-reported outcomes on pain, bodily functions, quality of life, cognitive function, and level of physical activity, along blood and faecal analyses, radiological changes and health economic analyses.

Statistical Considerations and Sample Size Calculation

The study is planned with an adaptive design, with an interim analysis after 50 participants. A team comprising a statistician and two scientists, including at least one clinician experienced in RCTs, will assess the primary outcome at six months. The analysis will be blinded to group identities and will determine the intervention's effect size. The results will guide on whether to adjust the sample size or intervention, especially if effects are smaller than expected.

Lacking prior data on this new physical activity intervention, we set an initial sample size aiming for a 50% improvement in severe sitting and walking difficulties in the intervention group compared to controls. Based on prior findings showing 30% prevalence of such issues and calculated with 80% power and a significance level of p<0.05, the required sample size was 121 patients per group. To account for non-compliance, 29 additional patients per group were added, resulting in a total of 300 participants, split evenly between the two groups.

Data Collection

Objective data to assess physical strength etc will be collected at baseline, at 6 and 12 months postoperatively. Patient reported data will be collected using a combination of online and paper-based methods. Baseline data will be collected at diagnosis with follow-up questionnaires administered at 6, 12, and 24 months post-surgery. These will cover aspects from socio-economic status to pain, quality of life, and kinesophobia. The tools will include established instruments like KASAM and custom scales derived through clinimetric methods (face-validated). Clinical data will be collected through national registers.

Data Analyses and Statistical Methods

Primary analyses will employ intention-to-treat approach, corrected for stratification variables and potential confounders. Descriptive statistics will summarize baseline characteristics, with inferential statistics (e.g., chi-squared tests, ANOVA) applied to primary and secondary outcomes. Multivariate regression analyses will explore predictors of successful outcomes, and health economic evaluations will assess cost-effectiveness.

External validity All patients with rectal cancer to be treated by abdominoperineal excision will be registered in the "screening log", including patients who do not meet the inclusion criteria, patients excluded after randomization, patients not giving consent to participation as well as those missed. All should be registered concerning date of diagnosis, sex, age, ASA class, cTNM, neoadjuvant treatment yes/no, type of operation/s. The reason for non-inclusion or exclusion will be noted.

Registration The trial is registered at ClinicalTrials.gov (No. [XXXX]) ensuring transparency and adherence to international standards.

Ethical Approval Ethical approval has been secured in Sweden (Swedish Ethical Board Authority approval No. 2024-08611-01) Informed consent will be obtained, respecting participant autonomy and confidentiality. The trial will be conducted according to the Helsinki declaration.

Timeline

1. Months 0-6: Finalize protocol, obtain ethical approval, and begin recruiting participants.
2. Months 7-18: Continue recruitment, involve more centers, initiate intervention, and collect baseline data and begin follow-up data collection.
3. Months 19-36: Complete intervention, conduct interim analyses, and begin follow-up data collection.
4. Months 37-48: Data collection outcome at 6 months, comprehensive data analysis, and dissemination of results. Follow up data collection.
5. Months 49-72: Data collection for outcome at 12 and 24 months, comprehensive data analysis, and dissemination of results

Clinical Relevance

The trial is clinically significant as it addresses the unmet need for effective postoperative rehabilitation in rectal cancer patients undergoing abdominoperineal excision (APE). This surgery, while necessary, leads to chronic mobility issues, such as sitting and walking difficulties, in up to 30% of patients, affecting their quality of life as well as activities of daily life. Standard postoperative care, which follows general physical activity guidelines, may not sufficiently address these challenges.

The trial evaluates a targeted exercise program designed to enhance muscle strength and balance. By doing so, it aims to directly address the mobility issues faced by patients post- surgery. If our hypothesis is correct, implementation of more effective rehabilitation strategies, improving functional outcomes and overall patient well-being should follow.

Additionally, by integrating health economic analyses we assess the cost-effectiveness of the intervention.

Preliminary Results

Unpublished (accepted in Diseases of the Colon and Rectum) data from our previous study comparing difficulties sitting and walking after APE versus anterior resection shows that this is much more frequent after APE and we therefore only include theese patients in the WASA-study.

Feasibility and Infrastructure

Feasibility The trial is coordinated by the Scandinavian Surgical Outcomes Research Group SSORG.The steering committee consists of experienced researchers with extensive knowledge in clinical RCT studies. There is a well established structure for managing recruitment and data. Data retrieval, management and analyses will be conducted using secure platforms (e.g., REDCap), ensuring high data integrity and participant privacy. Collaboration with other participating hospitals is established.

Infrastructure The Scandinavian Surgical Outcomes Research Group SSORG - established in 2009 at Sahlgrenska University Hospital is led by Professor Eva Haglind together with Professor Eva Angenete, who with associate professor Jennifer Park, me and two other post-docs constitute the senior researchers. Five PhD students are part of the group. Moreover there are three research nurses, a study administrator, one data manager (50 %) and two statisticians (80%). Collaborations frequently occur with other hospitals and regions, and the close cooperation with two university hospitals in Denmark have been ongoing since SSORg was established.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rectal cancer to be treated with/without neoadjuvant (chemo)radiation and abdominoperineal excision with or without mesh (APE/ELAPE) Informed consent Able to read and understand Swedish or Danish

Exclusion Criteria:

* Patients with rectal cancer to be operated by extended abdominoperineal excision (ELAPE) requiring musculocutaneous or muscular flaps to be operated by Hartmann's procedure to be operated by anterior resection (low or high) participation in other randomized trials in conflict with the protocol and endpoints of the WASA trial Not understanding Swedish or Danish Patients reporting habit of physical activity exceeding the WHO-recommendations (150 min + two strength sessions) at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2031-04-01 (Estimated)

PRIMARY OUTCOMES:
Can a specific physical online training program decrease sitting and walking difficulties 12 months after abdominoperineal excision for rectal cancer compared with standard care (self-administered aerobic training according to WHO recommendations only)? | 12 months
  Patient reported sitting and walking difficulties by validated questions in questionnaire with items from "no difficulties" to "severe difficulties".

SECONDARY OUTCOMES:
Self-reported problems with sitting and/or walking and physical activity | 6 and 24 months
  Patient reported sitting and walking difficulties by validated question in questionnaire at 6 and 24 months with items from "no difficulties" to "severe difficulties"
Objective tests | baseline, 6, 12 and 24 months
  Balance test as time in seconds standing on one leg, measured by a research nurse
Pain | 6, 12 and 24 months
  Pain, as reported by patient using validated instrument, Body Pain Inventory - Short Form (BPI-SF) included in questionnaire. Scored 0 (no pain) -10 (worst) on up to seven items.
Comprehensive Complication Index (CCI) | Within 30 and 90 days of abdominoperineal excision surgery
  Postoperative complications classified by CCI. Each complications is graded by Clavien-Dindo system and added into a score from 0 (no complications) to 100 (death).
Re-admissions | Within 12 and 24 months of abdominoperineal excision surgery
  Readmissions retrieved from hospital records, number of occasion
Parastomal hernia | 12 months after abdominoperineal excision surgery
  Retrieved by clinical record form, at clinical examination and radiology
Length of hospital stay | within 12 months and 24 months of abdominoperineal excision surgery
  Total length of hospital stay in days, retrieved from hospital records
Mortality | 30 days, 1, 2 and 5 years
  Retrieved from the Swedish/Danish National Cause of Death Register, date and cause of death
Health economic analysis | 24 months after abdominoperineal excision surgery
  Using data collected in the trial adding registered clinical costs, from health care cost-register in Sweden (KKP-register) with sensitivity analyses.
Perineal hernia | 12 months after abdominoperineal excision surgery
  Diagnosed through CT/MRI of the pelvic region
Biomarkers | Baseline, 4 weeks and 12 months
  Blood sample analyzed for markers for inflammation, such as inflammatory proteins
Faecal sample | baseline, 4 weeks and 12 months
  Analysis of kalprotectin and microbiome in faeces
Cognition | baseline, 6,12 and 24 months after abdominoperineal excision surgery
  Measured by specific questions on memory function in SF 36 instrument, items ranging from "no (problems)" to "more than 3 times per day"
Fatigue | 6, 12 and 24 months
  Measured by specific questions in SF 36
Activities of daily life | baseline, 6,12 and 24 months
  Measured by specific questions in EQ5D with items raning from "no (problems)" to "cannot perform activity"
Bodily functions | baseline, 6, 12 and 24 months
  Measured by validated questions in questionnaire, no score involved. Items ranging from "no problem" to "problem at least 1 time per day"
Quality of life | 6,12 and 24 months
  Quality of life as reported by patient validated question in questionnaire: "How would you describe your quality of life during the last month" answered in a 7 point Likert scale from "worst possible" to "best possible"
Muscle thickness | 12 months
  Diagnosed through CT/MRI of the buttocks/pelvic region
Fibrosis in pelvic region | 12 months
  diagnosed through CT/MRI of the pelvic region
Degree pf physical activity | 6,12 and 24 months
  PAtient reported by specific question (Saltin-Grimby) in questionnaire
Health economic analysis | 24 months
  comparison of intervention vs control by costs of intervention (one group), costs of hospital care, costs of sick-leave, using health economic models and sensitivity analsyes
Microbiota | 6 months
  determined in faecal sample
From sitting to standing | baseline, 6, 12 and 24 months
  Number of times rising from sitting to standing position during 30 seconds, measured by a research nurse
Walk test | baseline, 6, 12 and 24 months
  Time to walk 10 meters, measured by a research nurse
Grip strength | baseline, 6 and 12 months
  Hand grip strength tested by dynamometer, measured in kg by a research nurse
Reoperation | Within 12 and 24 months after abdoinomperineal escision surgery
  Retrieved from hospital records and described by type of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Charlotta E Larsson, MD, PhD, Principal Investigator — Department of Surgery, SSORG - Scandinavian Surgical Outcomes Research Group, Institute of Clinical Sciences, Sahlgrenska Academy, University of Gothenburg, Gothenburg, Sweden and Region Västra Götaland, Sahlgrenska University Hospital Östra
Locations (1):
- Department of Surgery, SSORG - Scandinavian Surgical Outcomes Research Group, Institute of Clinical Sciences, Sahlgrenska Academy, University of Gothenburg, 416 85 Gothenburg, Sweden., Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahmoudian A, Lohmander LS, Dahlberg LE, Kiadaliri A. Digital Self-management, Analgesic Use, and Patient-Reported Outcomes in Knee or Hip Osteoarthritis. Arch Phys Med Rehabil. 2024 Oct;105(10):1821-1828. doi: 10.1016/j.apmr.2024.05.033. Epub 2024 Jun 10. PMID 38866226
- [Background] Onerup A, Andersson J, Angenete E, Bock D, Borjesson M, Ehrencrona C, Fagevik Olsen M, Larsson PA, de la Croix H, Wedin A, Haglind E. Effect of Short-term Homebased Pre- and Postoperative Exercise on Recovery After Colorectal Cancer Surgery (PHYSSURG-C): A Randomized Clinical Trial. Ann Surg. 2022 Mar 1;275(3):448-455. doi: 10.1097/SLA.0000000000004901. PMID 33843798
- [Background] Onerup A, Angenete E, Bonfre P, Borjesson M, Haglind E, Wessman C, Nilsson H. Self-assessed preoperative level of habitual physical activity predicted postoperative complications after colorectal cancer surgery: A prospective observational cohort study. Eur J Surg Oncol. 2019 Nov;45(11):2045-2051. doi: 10.1016/j.ejso.2019.06.019. Epub 2019 Jun 12. PMID 31217078
- [Background] https://iris.who.int/bitstream/handle/10665/44399/9789241599979_eng.pdf?seque nce=1 2019 Nov;45(11):2045-2051.
- [Background] Bjorklund Sand L, Larsson C, Gronkvist R, Haglind E, Angenete E. Persistent Sitting and Walking Difficulties After Abdominoperineal Excision and Anterior Resection: Results From the Quality of Life in Rectal Cancer Study. Dis Colon Rectum. 2025 Jun 1;68(6):704-712. doi: 10.1097/DCR.0000000000003710. Epub 2025 Mar 14. PMID 40085057
- [Background] Asplund D, Prytz M, Bock D, Haglind E, Angenete E. Persistent perineal morbidity is common following abdominoperineal excision for rectal cancer. Int J Colorectal Dis. 2015 Nov;30(11):1563-70. doi: 10.1007/s00384-015-2328-1. Epub 2015 Aug 6. PMID 26245948